CLINICAL TRIAL: NCT01563705
Title: Prospective Follow-up of Patients With Glycogen Storage Disease Type III
Acronym: PRO GSDIII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-A00615-34
Record Dates: First submitted 2012-03-21; First posted 2012-03-27 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Neuromuscular Disorders
Keywords: Neuromuscular Disorders; GSD III; glycogen storage disease
MeSH Terms: conditions — Neuromuscular Diseases; Glycogen Storage Disease Type III; Glycogen Storage Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Different motor function tests — Time to rise from a chair, time to go from lying to sitting, time to go from lying to standing, time to cover 10 meters, time to climb 4 steps
Procedure: Manual dexterity assessment — Purdue pegboard test

SUMMARY:
The aim of this study is to improve knowledge of natural history and methods of monitoring the evolution of Glycogen storage disease type III regarding the muscle and to study the prospective approach of large series of patients, and using the same protocol for the follow up of the children and adults.

ELIGIBILITY:
Inclusion Criteria:

* patients with a debranching enzyme deficiency confirmed by enzymatic analysis (debranching enzyme deficiency).
* Written consent
* Age: at least 10 years
* Affiliated with a social security system

Exclusion Criteria:

* Pregnant and lactating women

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Knee flexion and extension strength | at baseline
Knee flexion and extension strength | 2 years after baseline
Knee flexion and extension strength | 4 years after baseline
Time to perform each motor function test | at baseline
Time to perform each motor function test | 2 years after baseline
Time to perform each motor function test | 4 years after baseline
Gait speed measured during the 6 minutes walk test | at baseline
Gait speed measured during the 6 minutes walk test | 2 years after baseline
Gait speed measured during the 6 minutes walk test | 4 years after baseline

SECONDARY OUTCOMES:
Accelerometric variables measured for the 6 minutes walk test | At baseline
Accelerometric variables measured for the 6 minutes walk test | 2 years after baseline
Accelerometric variables measured for the 6 minutes walk test | 4 years after baseline
NMR variables measured during each specific NMR sequence | at baseline
NMR variables measured during each specific NMR sequence | 2 years after baseline
NMR variables measured during each specific NMR sequence | 4 years after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Myologie, Paris, France